CLINICAL TRIAL: NCT04071275
Title: Does Transcranial Direct Current Stimulation (tDCS) Improve the Effect of Mirror Therapy? A Double-blind Randomized Controlled Study in Patients With Phantom Limb Pain.
Brief Title: Assessing Possible Additive Effects of tDCS and Mirror Therapy Treatments for Phantom Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, Hagay Amir, Medical Diractor, Loewenstein Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOH_3107-2018-003552
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Phantom Limb Pain
MeSH Terms: conditions — Phantom Limb | interventions — Transcranial Direct Current Stimulation; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mirror therapy (Active Comparator): Subjects will be asked to perform specific movements (using the unaffected limb while watching its mirrored reflection for 20 minutes per day, for 10 treatment days, completed during two weeks (every weekday, excluding weekends)
  Interventions: Other: Mirror therapy
- Mirror therapy + sham tDCS (Sham Comparator): Subject will undergo the mirror therapy treatment, as in the first study arm. In addition, at the same time, a sham tDCS treatment will be applied.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Other: Mirror therapy
- Mirror therapy + active tDCS (Experimental): Subject will undergo the mirror therapy treatment, as in the first study arm. In addition, at the same time, an active tDCS treatment will be applied.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS); Other: Mirror therapy

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — tDCS is a non-invasive technique that allow the administration of low currents directly to the scalp. The currents affect the cortex, and result in changes to the membrane potential of neurons in the stimulated area. This in turn affects the tendency of those neurons to generate action potentials.
  Arms: Mirror therapy + active tDCS; Mirror therapy + sham tDCS
Other: Mirror therapy — Mirror therapy is a behavioral technique that proven useful for the treatment of phantom pain, yet the analgesic effects are unfortunately moderate and not long lasting. The assumed underlying mechanism of mirror therapy treatment is the induction of neuronal plasticity in the opposite direction than the abnormal reorganization of the cortex (due to the amputation), and by that relive pain.

SUMMARY:
In this study we will examine assess if treatment with transcranial Direct Current Stimulation (tDCS) improve the analgesic effects of mirror therapy for patients with phantom pain of lower extremity. The study will include 3 arms: only mirror therapy, mirror therapy + sham tDCS, and mirror therapy + active tDCS.

DETAILED DESCRIPTION:
Phantom pain following amputation is difficult to treat, resulting in many patients who suffer. One of the mechanisms suspected to contribute to phantom pain is abnormal plasticity and reorganization of the cortex.

Mirror therapy is a behavioral technique that proven useful for the treatment of phantom pain, yet the analgesic effects are unfortunately moderate and not long lasting. The assumed underlying mechanism of mirror therapy treatment is the induction of neuronal plasticity in the opposite direction than the abnormal reorganization of the cortex (due to the amputation), and by that relive pain.

tDCS is a non-invasive technique that allow the administration of low currents directly to the scalp. The currents affect the cortex, and result in changes to the membrane potential of neurons in the stimulated area. This in turn affects the tendency of those neurons to generate action potentials.

It was hypothesize that combination of mirror therapy and tDCS treatment could result in additive effects. According to this hypothesis, the effects of the mirror therapy could be enhanced by the tDCS treatment. The aim of the current study is to investigate this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Underwent unilateral lower limb amputation in the past 3 months. A
3. Reported average phantom pain of 4 or more in the past week.
4. No change in other medications 1 week prior to enrollment, not including SOS.
5. Able understand the purpose of the study and to provide informed consent.

Exclusion Criteria:

1. Ferromagnetic metal in the head or neck.

1. Epilepsy or prior seizures within the last 1 year.
2. Suffering from severe depression
3. History of unexplained fainting or loss of consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-22 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) | between baseline week and 4 weeks after the end of the treatment
  The Visual Analog Scale (VAS) of the average Phantom Limb Pain in the past week will serve as primary measure. The primary outcome is the changes in the VAS score between baseline week and 4 weeks after the end of the treatment. VAS is a widely used, continuous measure of pain intensity, with scores ranging between 0-10, higher scores reflecting higher pain intensity.

SECONDARY OUTCOMES:
McGill total score | between baseline week and 4 weeks after the end of the treatment
  Changes in short-form McGill total score between baseline week and 4 weeks after the end of the treatment. The McGill Pain Questionnaire (MPQ) is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is composed of 78 words, of which respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word. The short-form McGill Pain Questionnaire (SF-MPQ) is a shorter version of the original MPQ. The pain rating index has 2 subscales: 1. Sensory subscale with 11 words, and 2. Affective subscale with 4 words from the original MPQ. These words or items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe. There's also one item for present pain intensity.
McGill sensory sub-score | between baseline week and 4 weeks after the end of the treatment
  Changes in short-form McGill sensory sub-score between baseline week and 4 weeks after the end of the treatment. The McGill Pain Questionnaire (MPQ) is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is composed of 78 words, of which respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word. The short-form McGill Pain Questionnaire (SF-MPQ) is a shorter version of the original MPQ. The pain rating index has 2 subscales: 1. Sensory subscale with 11 words, and 2. Affective subscale with 4 words from the original MPQ. These words or items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe. There's also one item for present pain intensity.
Changes in the worst pain | between baseline week and 4 weeks after the end of the treatment
  Changes in the worst pain over the past week (taken from the Brief Pain Inventory (BPI questionnaire) between baseline week and 4 weeks after the end of the treatment. The scale rapidly assesses the severity of pain and its impact on functioning. No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.
Changes in the average pain | between baseline week and 4 weeks after the end of the treatment
  Changes in the average pain over the past week (taken from the Brief Pain Inventory (BPI questionnaire) between baseline week and 4 weeks after the end of the treatment. The scale rapidly assesses the severity of pain and its impact on functioning. No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.
Changes in the VAS score | between baseline week and 12 weeks after the end of the treatment
  Changes in the VAS score between baseline week and 12 weeks after the end of the treatment. VAS is a widely used, continuous measure of pain intensity, with scores ranging between 0-10, higher scores reflecting higher pain intensity.
Changes in short-form McGill total score | between baseline week and 12 weeks after the end of the treatment
  Changes in short-form McGill total score between baseline week and 12 weeks after the end of the treatment. The McGill Pain Questionnaire (MPQ) is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is composed of 78 words, of which respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word. The short-form McGill Pain Questionnaire (SF-MPQ) is a shorter version of the original MPQ. The pain rating index has 2 subscales: 1. Sensory subscale with 11 words, and 2. Affective subscale with 4 words from the original MPQ. These words or items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe. There's also one item for present pain intensity.
Changes in short-form McGill sensory sub-score | between baseline week and 12 weeks after the end of the treatment
  Changes in short-form McGill sensory sub-score between baseline week and 12 weeks after the end of the treatment. The McGill Pain Questionnaire (MPQ) is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is composed of 78 words, of which respondents choose those that best describe their experience of pain. Scores are tabulated by summing values associated with each word. The short-form McGill Pain Questionnaire (SF-MPQ) is a shorter version of the original MPQ. The pain rating index has 2 subscales: 1. Sensory subscale with 11 words, and 2. Affective subscale with 4 words from the original MPQ. These words or items are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate and 3 = severe. There's also one item for present pain intensity.
Changes in the worst pain | between baseline week and 12 weeks after the end of the treatment
  Changes in the worst pain over the past week (taken from the Brief Pain Inventory (BPI questionnaire) between baseline week and 12 weeks after the end of the treatment. The scale rapidly assesses the severity of pain and its impact on functioning. No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.
Changes in the average pain | between baseline week and 12 weeks after the end of the treatment
  Changes in the average pain over the past week (taken from the Brief Pain Inventory (BPI questionnaire) between baseline week and 12 weeks after the end of the treatment. The scale rapidly assesses the severity of pain and its impact on functioning. No scoring algorithm, but "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference.

CONTACTS AND LOCATIONS:
Overall Officials: Nitza Segal, M.A, Study Chair — Leowenstein Hospital
Locations (1):
- Loewenstein Hospital, Raanana, Israel

IPD SHARING:
Plan to Share IPD: No